CLINICAL TRIAL: NCT05554809
Title: Crossover-effect of Unilateral Dynamic Versus Static Stretch of Hamstrings Muscle on Hamstrings Muscle Length - a Randomized Controlled Trial
Brief Title: Unilateral Stretch Crossover Effect RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Luleå Tekniska Universitet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LuleaTU
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Muscle Tightness; Stretch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor are not aware of the participants group allocation at time of measurement of outcome measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dynamic stretching (Experimental)
  Interventions: Other: Strecthing
- Static stretching (Experimental)
  Interventions: Other: Strecthing
- Controll (Active Comparator)
  Interventions: Other: Strecthing

INTERVENTIONS:
Other: Strecthing — Comparing the crossover-effect of dynamic versus static stretching

SUMMARY:
The crossover-effect within resistance- and strength training is more or less confirmed with multiple studies showing similar results. The studies shows an increase in muscle strength within the contralateral extremity being exercised. Regarding muscle length or mobility (flexibility) the crossover-effect have not been studied.

For a person to gain an increase in muscle strength mobility training in the form of stretching and flexibility training of our skeletal muscle is a common exercise. However, the evidence are scare and there are only a few studies comparing the effect of prolonged static stretching (> 90 sec) and dynamic flexibility training as to which of these methods has the best length-enhancing effect over time.

The purpose of this study is to compare the crossover-effect of eight weeks of oneleg dynamic flexibility training versus oneleg prolonged static stretching versus a nonstretching controlgroup on mobility in the hamstring muscles in adults with reduced mobility of the hamstring muscle. The aim is also to compare the sustained effect of flexibility training between the two groups, eight weeks after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Passiv straigth leg raise < 70 degrees
* Read and understand swedish

Exclusion Criteria:

* Injuries within the hamstrings muscle past 3 month
* Disabilities within the muscloskeletal system (i.e. lower back, thoracic spine, cervikal spine, hip, knee, ankle, fot) affecting the participants life
* Neurological, inflammatoric or heart-diseases
* Nociplasic pain disorders
* Medication with possibility affecting muscle strength of flexibility
* Positive neurodynamic test of the lower extremity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Passiv straigth leg raising | 5 minutes
  Muscle length of the hamstrings muscle will be measured via degress of hip flexion at a passive straigth leg raise of the lower extremity. One leg at a time.
Active knee extension | 5 minutes
  The person will lay supine with a 90 degress of hip flexion towards a bar against the thigh. Thereafter the person will perform an active knee extensor as far as possible and the degrees of kneeflexion will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Luleå university of Technology, Luleå, Norrbotten County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided